CLINICAL TRIAL: NCT04715178
Title: Specimen Banking With Clinical and Genomic Data Registry With the Establishment of Tumor Models for Pediatric Cancers
Brief Title: Beat Childhood Cancer Specimen Banking and Data Registry
Status: Recruiting | Type: Observational
Sponsor: Giselle Sholler (Other)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Beat Childhood Cancer Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Other Study IDs: BCC-BIO-001
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Cancer; Survivorship
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — whole blood, serum, urine, bone marrow, CSF, bucal swabs, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected or confirmed pediatric solid tumors: Patients with suspected or confirmed pediatric solid tumors
  Interventions: Other: No intervention- registry only

INTERVENTIONS:
Other: No intervention- registry only — No intervention- registry only

SUMMARY:
This is an observational data registry study of pediatric cancer patients at participating Beat Childhood Cancer Consortium sites involving specimen banking and data collection.

DETAILED DESCRIPTION:
This observational registry and banking study is being performed on a large cohort of subjects who have received molecular testing to better understand the relationship between genomic and molecular information and clinical outcomes, and to enable timely and informed treatment decisions by physicians for their cancers. We hypothesize that large gene panels, sequencing (DNA/RNA), and epigenetics of tumors can identify molecular aberrations that can be leveraged to offer more effective treatment. Findings may highlight additional areas of research required to better understand the molecular underpinnings of the relationship between molecular abnormalities and disease. Banked specimens and the creation of tumor cell lines and xenograft models will facilitate further advancement of this research.

ELIGIBILITY:
Inclusion Criteria:

* No age restrictions
* Subjects that fit into one of the following categories:

  1. Subjects with suspected or confirmed cancers of childhood, adolescence, or young adulthood.
  2. Survivors of a cancer of childhood, adolescence, or young adulthood (> 6 months off last therapy for cancer)
  3. Subjects with a disease-matched condition
  4. Healthy volunteers- including any participants with medical conditions that are not disease-matched.
* Written informed consent in accordance with institutional and FDA guidelines must be obtained from all subjects (or subjects' legal representative).

Exclusion Criteria:

* Subject or his/her legally authorized representative (where applicable) did not consent for specimen banking and data collection for this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric cancer subjects, survivorship, and healthy volunteers at The Pennsylvania State University and participating Beat Childhood Cancer Research Consortium sites.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Create a data registry of clinical and molecular/genomic data | 10 Years
  Create a data registry of clinical and molecular/genomic data from cancer patients who have undergone biopsy or surgical resection for clinical care to better understand the relationship between genomic and molecular information and clinical outcomes.
Determine number and types of genomic alterations within tumor types/subtypes | 10 Years
  Define genomic landscape of pediatric cancers through the determination of the number and types of genomic alterations within tumor types/subtypes, across tumor types, and tumor evolution over time.
Evaluate the rate of actionable genomic alternations | 10 Years
  Evaluate the rate of actionable genomic alternations resulting in associated targeted therapies relative to all actionable genomic alterations.
Evaluate the correlation of baseline genomic alterations with clinical outcome. | 10 Years
  Evaluate the correlation of baseline genomic alterations with clinical outcome.
Identify biomarkers that predict risk of adverse outcomes that occur following pediatric cancer therapy. | 10 Years
  Identify biomarkers that predict risk of adverse outcomes that occur following pediatric cancer therapy.

SECONDARY OUTCOMES:
Bank additional specimens available for future research projects | 10 Years
  Bank additional specimens available for future research projects
Develop cell line and xenograft models of pediatric cancers for future research | 10 Years
  Develop cell line and xenograft models of pediatric cancers for future research
Identify biomarkers that predict risks of disease states in subject controls that did not receive cancer therapy. | 10 Years
  Identify biomarkers that predict risks of disease states in subject controls that did not receive cancer therapy.
Identify biomarkers that may predict risk of disease dependent on sex, race, ethnicity, or the presence of comorbidities. | 10 Years
  Identify biomarkers that may predict risk of disease dependent on sex, race, ethnicity, or the presence of comorbidities.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Sholler, MD, Study Chair — Beat Childhood Cancer
Locations (18):
- United States (18):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Rady Children's Hospital, San Diego, California
  - Connecticut Children's Hospital, Hartford, Connecticut
  - Nicklaus Children's Miami, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - Norton Children's Research Institute/Affiliated with University of Louisville School of Medicine, Louisville, Kentucky
  - Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Levine Children's Hospital, Charlotte, North Carolina
  - AH Wake Forest Baptist - Brenner Children's Hospital, Winston-Salem, North Carolina
  - Randall Children's Hospital, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center and Children's Hospital, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Dell Children's Blood and Cancer Center, Austin, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Beat Childhood Cancer Consortium website — https://research.beatcc.org/